CLINICAL TRIAL: NCT04941508
Title: Mother's Recorded Voice: a Neglected Therapeutic Stance for Pediatric Postoperative Agitation
Brief Title: Mother's Recorded Voice Versus Dexmedetomidine on Postoperative Agitation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Makram Soliman, Lecturer of anesthesia and ICU, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17300621
Record Dates: First submitted 2021-06-15; First posted 2021-06-28 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Agitation, Emergence
MeSH Terms: conditions — Emergence Delirium | interventions — Dexmedetomidine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mother's recorded voice (Experimental): Children will be exposed to the mother's voice.
  Interventions: Behavioral: the mother's recorded voice
- Dexmedetomidine IV (Experimental): Children will be given dexmedetomidine injection.
  Interventions: Drug: Dexmedetomidine
- Saline placebo IV (Placebo Comparator): Children will be given normal saline.
  Interventions: Other: saline 0.9% placebo

INTERVENTIONS:
Behavioral: the mother's recorded voice — Children will be assigned to listen to the mother's recorded voice at 2 times (in the holding area 3 minutes before induction of anesthesia till induction of anesthesia is ended) and (during emergence from anesthesia till complete recovery).
  Arms: Mother's recorded voice
Drug: Dexmedetomidine — Children will be given a single bolus of dexmedetomidine 0.2 µ/kg IV at 2 times (in the holding area 3 minutes before induction of anesthesia) and (at the end of surgery).
  Other Names: Precedex
  Arms: Dexmedetomidine IV
Other: saline 0.9% placebo — Children will be given the same volume of saline at 2 times (in the holding area 3 minutes before induction of anesthesia) and (at the end of surgery).
  Other Names: Normal saline
  Arms: Saline placebo IV

SUMMARY:
The aim of this study is to compare the efficacy of mother's recorded voice versus dexmedetomidine injection on postoperative agitation in children undergoing elective surgery.

DETAILED DESCRIPTION:
A written informed consent will be taken from the patients' legal guardians.Patients will be assigned randomly to three groups (30 subjects each) to be anesthetized and either randomly assigned to listen to the mother's recorded voice at 2 times (in the holding area 3 minutes before induction of anesthesia till induction of anesthesia is ended) and (during emergence from anesthesia till complete recovery) (Group M) or will be given a single bolus of dexmedetomidine 0.2 µ/kg IV at 2 times (in the holding area 3 minutes before induction of anesthesia) and (at the end of surgery) (Group D) or given the same volume of saline IV at 2 times (in the holding area 3 minutes before induction of anesthesia) and (at the end of surgery) (Group C).To keep blinding, group M will be injected IV with the same volume of saline at the same 2 times as in groups D & C while in groups D & C, headphones will be putted as in group M at the same 2 times with no recorded voice.

ELIGIBILITY:
Inclusion Criteria:

* Children (age 4-9 years)
* American Society of Anesthesiologists physical status (ASA) I-II who will be listed for outpatient elective surgery under general anesthesia.

Exclusion Criteria:

* Developmental delays
* Neurological diseases
* Deafness
* Hearing impairment
* Maternal mutism
* Absence of the mother

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2021-11-05 (Actual)

PRIMARY OUTCOMES:
Pediatric anesthesia of emergence delirium (PAED) score | 2 hours Postoperative
  Emergence delirium (ED) will be measured by the pediatric anesthesia of emergence delirium (PAED).The scores for each of the five listed behaviours(makes eye contact with caregiver, actions are purposeful,aware of surroundings, restless and inconsolable) are added to achieve a total score (maximum score of 20). A score of >12 yields 100% sensitivity and 94.5% specificity for the diagnosis of ED

SECONDARY OUTCOMES:
Face, Legs, Activity, Cry, and Consolability (FLACC) score | 24 hours Postoperative
  Pain will be measured by Face, Legs, Activity, Cry, and Consolability (FLACC) score ranging from 0 to 10 where 0= relaxed and no pain, 1-3= mild pain/discomfort, 4-6= moderate pain, 7-10= severe discomfort/pain.

CONTACTS AND LOCATIONS:
Overall Officials: Omar Soliman, MD, Study Director — Assiut University
Locations (2):
- Egypt (2):
  - Assiut university hospital, Asyut
  - Omar Soliman, Asyut

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Manyande A, Cyna AM, Yip P, Chooi C, Middleton P. Non-pharmacological interventions for assisting the induction of anaesthesia in children. Cochrane Database Syst Rev. 2015 Jul 14;2015(7):CD006447. doi: 10.1002/14651858.CD006447.pub3. PMID 26171895